CLINICAL TRIAL: NCT06053034
Title: Assessing the Effectiveness of the Solio Alfa Cure Plus Device in Treating Low Back Pain: a Randomized Controlled Study
Brief Title: Effectiveness of the Solio Alfa Care Plus Device in Treating Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Itay GoorAryeh, Head of Pain Clinic, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 847521SMC
Record Dates: First submitted 2023-09-10; First posted 2023-09-25 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sham device (Sham Comparator): a round device equipped with a strap for hand holding, it is to be used while connected to a socket. The device is used by an assistant (usually a family member) on the participant's back for 20 minutes while moving it around in circles on the lower back.
  Interventions: Device: Solio alpha cure plus
- Solio Alpha Plus (Active Comparator): The SOLIO Alfa Cure Plus Device for patients with LBP- is a round device equipped with a strap for hand holding, it is to be used while connected to a socket. The device is used by an assistant (usually a family member) on the participant's back for 20 minutes while moving it around in circles on the lower back. It should be mentioned this is the first trial in Home-RF using an external
  Interventions: Device: Solio alpha cure plus

INTERVENTIONS:
Device: Solio alpha cure plus — The SOLIO Alfa Cure Plus is the only home-use device with FDA clearance that uses the proprietary synergy of three energy sources (IR, RF, and LLLT), and this study aims to assess the SOLIO Alfa Cure Plus's efficiency in providing pain relief. This technology is the first noninvasive and patented home RF device. SOLIO Alfa Cure Plus uses continuous RF, the internal controller reduces the RF power while reaching the treatment temperature of 39- 42 Celsius.The SOLIO Alfa Cure Plus Device is a round device equipped with a strap for hand holding, it is to be used while connected to a socket. The device is used by an assistant (usually a family member) on the participant's back for 20 minutes while moving it around in circles on the lower back.

SUMMARY:
Objectives: This double-blind, randomized, prospective, single-centre study evaluated the effectiveness of radiofrequency therapy by the SOLIO Alfa Cure Plus in the treatment of a non-specific low back pain (LBP) Methods: Thirty-seven patients completed pain, disability, and lower back flexibility scales. Randomization was obtained by having an equal amount of sham and real devices and distributing them randomly to patients out of a box where the devices were.

DETAILED DESCRIPTION:
Studies have shown that some generally recommended first-line medications for low back pain (LPB) are only slightly more effective than placebo controls in double-blind randomized trials [10]. For instance, physical exercise in combination with manual therapy often produces short-term results [15], such as the epidural corticosteroid injection that presents a complication rate between 0% and 9.65%. At the same time, various energy sources are thought to have great potential for both general healing and pain relief [11] [12] and there are several available devices that make use of this technology [13].

Infrared therapy (IR) can reach muscles, nerves and even bones, where it reduces inflammation by accessing inner layers of tissues. The use of IR therapy has been shown to accelerate wound healing, ease arthritis knee pain, increase endorphin levels, and activate neuromodulators [19] without any side effects. According to a recent study, IR therapy is beneficial for chronic non-specific LBP sufferers in terms of comfort, function, lumbar range of motion, and back extensor endurance [20].

Radio frequency (RF) therapy shows promise as a healing strategy in a variety of etiologies [22]- [24] and it one of the most common energy sources for producing therapeutic heat levels. RF energy is delivered to soft tissue as part of the mechanism's biophysical therapeutic mode to relieve pain, as well as enhancing collagen formation, vascularization, and collagen structure in the tissue [22]- [24]. Another energy source is the tow-level laser treatment (LLLT), known to induce analgesia, reduce inflammation, and promote healing in a variety of musculoskeletal diseases. This technique is based on the theory that light causes biochemical changes in cells like photosynthesis in plants. [26]. LLLT may also be used as an adjuvant therapy for pain management in patients with neurologic impairments and neuropathic pain [27].

The techniques are potential tools for controlling pain in a variety of etiologies, but additional research appears to be needed to fully develop the therapeutic and mechanistic role of these techniques. No device combining all three approaches has ever been objectively assessed in a randomized clinical trial for pain management. The SOLIO Alfa Cure Plus is the only home-use device with FDA clearance that uses the proprietary synergy of three energy sources (IR, RF, and LLLT), and this study aims to assess the SOLIO Alfa Cure Plus's efficiency in providing pain relief. This technology is the first non-invasive and patented home RF device. SOLIO Alfa Cure Plus uses continuous RF, the internal controller reduces the RF power while reaching the treatment temperature of 39- 42 Celsius.

These three treatment modalities are hypothesized to affect the physiological issue at many levels, causing tissue regeneration and pain relief at the cellular and tissue levels, as well as changing sensory nerves and cell molecular makeup [18], [20], [25], [27]. Our goal was to determine whether the RF component of the treatment has an effect on back pain relief.

ELIGIBILITY:
Inclusion Criteria:

* Patients with LBP lasting 6 weeks and less than 6 months (NRS) of 4 or higher), between 18 to 70 years old that possessed assistance of family members

Exclusion Criteria:

* patients with fibromyalgia, pregnancy, pacemaker implant, hyper coagulation, cognitive impairment, psychosis diagnosis, addiction, opiate usage, malignant cancer, and BMI > 35 or 18.5

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 1 month
  The Pain Numerical Rating Scale (NRS) - it is an 11-point scale for self-report of pain. It is the most commonly used unidimensional pain scale. The respondent selects a whole number (integers 0-10) that best reflects the intensity (or other quality if requested of his/her pain

SECONDARY OUTCOMES:
Disability score | 1 month
  10 questions about the participant's daily experience with their back pain and how it affects diverse day to day activities (e.g., social life, work life, walking and standing, etc.).

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel

IPD SHARING:
Plan to Share IPD: Undecided